CLINICAL TRIAL: NCT03471533
Title: Clinical Trial and Randomized Efficacy of a Natural Ingredient on the Arterial Tension of Normother Subjects or With Arterial Hypertension Grade i Without Pharmacological Treatment
Brief Title: Efficacy of a Natural Ingredient on Blood Pressure
Acronym: FISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UCAM-CFE-0001
Record Dates: First submitted 2018-02-27; First posted 2018-03-20 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial, with two parallel branches, (experimental product and placebo), double blind and unicentric.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ëxperimental (Experimental): Consumption during 84 days of Lippia citriodora 325 mg + Hibiscus sabdariffa 175 mg.
  Two capsules a day will be consumed thirty minutes before breakfast for 84 days.
  Interventions: Dietary Supplement: nutraceutical: experimental product
- Placebo (Placebo Comparator): Consumption during 84 days of saccharose. Two capsules a day will be consumed thirty minutes before breakfast for 84 days.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: nutraceutical: experimental product — 84 days of consumption
  Arms: Ëxperimental
Dietary Supplement: placebo — 84 days of consumption
  Arms: Placebo

SUMMARY:
Randomized controlled trial with two parallel branches (experimental product and placebo), double blind and unicentric with which it is intended to evaluate the efficacy of the product under investigation against placebo on blood pressure of normotensive subjects or with hypertension grade I without Pharmacotherapy. The subjects that meet the selection criteria will make a total of five visits to the research laboratory and perform the tests that were pre-established in the protocol. Later, a statistical analysis will be carried out with the variables measured in the study to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes between 18-65 years old.
* Systolic blood pressure between 120 and 159 mmHg or diastolic blood pressure between 80 and 100 mm Hg. taken in basal conditions.
* Volunteers able to understand the clinical study and willing to comply with the procedures and requirements of the study

Exclusion Criteria:

* In pharmacological treatment of arterial hypertension.
* Subjects with acute diseases.
* Volunteers with a history or presence of chronic pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunological, dermatological, urological, neurological, psychiatric, cardiovascular or pathological conditions or malignant tumor disease that can modify the blood pressure of subjects.
* Subjected to major surgery in the last 3 months.
* Subjects who stopped smoking in the last 6 months or who intend to quit during the study.
* Subjects with allergies or eating disorders.
* Participation in another study that includes blood extractions or dietary intervention.
* Pregnant woman.
* Subjects whose condition does not make them eligible for the study, according to the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Assessing a change of blood pressure five times | Blood pressure measurements will be taken with a Holter on five separate occasions and for 24 hours each day. The measurements will be made at baseline and at 14, 28, 56 and 84 days of consumption of the product.
  blood pressure is measured with a holter

SECONDARY OUTCOMES:
body composition | Two densitometries will be performed. One at the beginning of the test, in basal conditions and another at the end of the test after 84 days of taking the product.e beginning and at the end
  Dual X-ray absorptiometry (DEXA)
body composition | A record of body composition will be made five times during the 84 days of consumption. Measures will be taken at baseline, at 14 days, 28, 56 and 84 days.
  Bioimpedancetry
blood samples | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of use.
  Glucidal metabolism and lipid metabolism. It was measured in milligrams per deciliter.
Subjective sensation of product consumption | Subjects will complete the hedonic scale four times. at 14, 28, 56 and 84 days of consumption of the product under study.
  5-point hedonic scale. There are five points, being 1 I do not like and 5 I like it a lot. A scale will be passed through paper.
physical activity | An accelerometer will be placed twice on the subjects. The first time at baseline and the second after taking 84 days of consumption of the product under study.
  accelerometer
Control of dietary intake | A nutritional registry will be carried out. The nutritional intake of for days in two periods will be collected. One record at the beginning and another at the end, that is, six days.
  Diet source
quality of life questionnaire | The cuestionnaire will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of use. The subjects have to answer 26 items on a scale of one to five, being one never and 5 always.
  questionnaire: WHOQOL-BREF
Gastrointestinal well-being evaluation | The questionnaire will be completed five times (GIQLI). It will be completed at baseline (without consumption of the product), at 14, 28, 56 and 84 days of consumption of the experimental product.
  Gastrointestinal quality of life questionnaire. The subjects have to answer 36 items on a scale of one to five, being 1 all the time and 5 never.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain